CLINICAL TRIAL: NCT05109078
Title: Single Dose Absorption, Distribution, Metabolism, and Excretion Study of [14C]- Rongliflozin in Healthy Male Participants
Brief Title: ADME Study of [14C]- Rongliflozin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DJT1116PG-DM-107
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]- Rongliflozin (Experimental): Patients will receive single dose of [14C]- Rongliflozin (Suspension, 50mg/100μCi)
  Interventions: Drug: [14C]- Rongliflozin

INTERVENTIONS:
Drug: [14C]- Rongliflozin — Patients will receive single dose of orally [14C]- Rongliflozin on Day 1

SUMMARY:
Study to Evaluate the Mass Balance and Biotransformation of Single Dose [14C]- Rongliflozin in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, 18 to 45 years at the time of screening.
2. Go to Weight>50 kg, Body mass index (BMI) is 19~26 kg/m2
3. Signing of informed consent
4. Participants are able to communicate well with the investigators and be able to complete the trial according to the Process.

Exclusion Criteria:

1. Physical examination, routine laboratory tests, 12-lead ECG, Chest X-ray, abdominal B-ultrasound, New Coronavirus Testing and other is abnormal and clinically significant.
2. Positive testing for HIV, HBsAg, HBeAb, HCVAb or Syphilis antibody.
3. CYP3A4, uridine diphosphoglucuronyl transferase(UGT) inducers or inhibitors, and P-gp, breast cancer resistance protein(BCRP) Substrates were taken within 28 days before screening.
4. Use of any prescription or over-the-counter drug, any vitamin product, health care drug or Chinese herbal medicine within 14 days prior to screening.
5. Participants who have participated in any clinical trials within 3 months prior to screening and have used thetest drug or medical devices.
6. Participants who have been vaccinated within 1 month before screening or plan to be vaccinated during the trial period.
7. A history of any clinically serious illness or condition, including but not limited to circulatory, endocrine, nervous,digestive, urinary, or blood, immune, mental, and metabolic diseases, that the investigator considers to be likely to affect the results of the study.
8. People who have had heart disease such as heart failure, angina pectoris, myocardial infarction, and clinically significant arrhythmia.
9. A history of urinary tract infection or repeated hypoglycemia.
10. Participants who had undergone major surgery or whose surgical incision was not completely healed within 6 months before the screening period;Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury.
11. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred withini 6 months before screening.
12. Significant clinical bleeding symptoms or definite bleeding tendency occurred within 3 months before screening.
13. Hemorrhoids or perianal diseases with regular/bleeding in the stool; Patients with gastrointestinal dysfunction, such as irritable bowel syndrome and inflammatory bowel disease, may be affected by drug absorption as determined by researchers.
14. Participants who have allergies or have special dietary requirements and cannot follow the standard diet.
15. Habitual constipation or diarrhea.
16. Heavy drinking or regular drinking in the six months preceding the screening period, or alcohol breath test results ≥20 mg/dL during the screening period.
17. Those who had smoked more than 5 cigarettes per day on average in the 3 months before the screening period or habitually used nicotine-containing products and were unable to quit during the test period.
18. Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.) in the 1 year prior to the screening period, or screening for positive urine drug abuse (drug) tests.
19. Habitual consumption of grapefruit juice or excessive consumption of tea, coffee and/or caffeinated beverages and failure to abstain during the study period.
20. Those with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection.
21. Workers engaged in conditions requiring long-term exposure to radioactivity; or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before the test or have participated inthe radiopharmaceutical labeling test.
22. Having family planning during the trial period and within 12 months after the last use of the drug, or not agreeing that subjects and their spouses should take strict contraceptive measures during the trial period and within 12 months after the last use of the drug.
23. Those who have lost blood or donated up to 400 mL within 3 months before the screening period, or those who have received blood transfusion, or those who plan to donate blood within 3 month after the end of this test.
24. As determined by the investigator, the subject has other factors that are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of 14C-labeled drug-related material (radioactivity in urine and fecal samples) | up to 14 days
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in urine and feces.
Identification of the Proportion of different metabolites to determine biotransformation pathway of Rongliflozin | up to 14 days
  Proportion of different metabolites(Rongliflozin and main metabolites).
Distribution of radioactivity in whole blood and plasma and the pharmacokinetics of total radioactivity in plasma | up to 11 days
  Radioactivity concentration in whole blood and plasma samples.

SECONDARY OUTCOMES:
Quantitive analysis of the concentrations of Rongliflozinand main metabolites in plasma using the validated liquid chromatography-tandem mass spectrometry(LC-MS/MS) to obtain pharmacokinetic data | up to 11 days
  The concentrations of Rongliflozin and main metabolites in plasma.
Adverse events | up to 21 days
  Adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China